CLINICAL TRIAL: NCT05394025
Title: COVID-19 Observational Research Collaboratory - Long-Term Outcomes (LTO) Study
Brief Title: COVID-19 Observational Research Collaboratory
Acronym: CORC LTO
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: C19 21-279
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: None Retained — No biospecimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Veterans who tested positive for COVID-19 (case): The investigators will organize the sampling of cases (and later of comparators) around the waves of the epidemic, as defined by their nadirs between national death rates-each approximately 3-4 months long. The investigators will initiate surveys of Veterans who have survived their initial SARS-CoV-2 infection. The viral infection "index date" will be defined as date of each patient's first positive test.
- Veterans who did not test positive for COVID-19 (comparator): To support causal inference, the investigators will also sample Veterans without COVID who are matched to participants with COVID-19. In general, cases will be compared to comparators matched on risk of developing COVID infection during a given wave.

SUMMARY:
This study aims to examine the long-term outcomes in Veterans infected and uninfected with SARS-CoV-2 using electronic health record information and structured surveys.

DETAILED DESCRIPTION:
Background: Early evidence suggests that the frequency and type of long term complications stemming from SARS-CoV-2 infection may depend on the severity of initial presentation. However, additional unidentified factors may also play a role including those related to the individual, the environment and/or the specific strain of the virus. The long-term health impacts of SARS-CoV-2 will have major implications for health care utilization, care processes and quality and costs of care for Veterans, both within the VA and in the community. Over 200,000 Veterans have had COVID-19. Although the long term consequences of this novel illness are unknown, it is clear they will often be significant. The overarching goal in the Long-Term Outcome Study (LTO) is to advance VA HSR&D research into the consequences and care of COVID-19 infection by developing and releasing integrated multi-modal data and results on long-term outcomes of COVID for use by VA clinical, research and operations communities. The investigators will do so via a coordinated program of data production and analysis using the VA electronic health record (EHR) and other administrative sources (e.g., Medicare), de novo longitudinal survey, and qualitative inquiry. This work will be closely coordinated with the COVID-19 Observational Research Collaboratory (CORC) Coordinating Center (CCC) and the burgeoning community of HSR&D-funded COVID researchers.

This study aims to examine the long-term outcomes in Veterans infected and uninfected with SARS-CoV-2.

Aim 1: Using VINCI-CDW data, patients will be identified who had a SARS-CoV-2 test since February 2020. The investigators will use a combination of traditional epidemiologic studies, and machine learning algorithms to determine the long term, multi-systemic and functional adverse outcomes and/or syndromes related to SARS-CoV-2. Members of the research team are currently developing methods to identify new onset and exacerbations in comorbidities following SARS-CoV-2 illness in Veterans.

Aim 2: Determine Veteran-Reported Outcome Effects Using Structured Survey on domains such as self- reported symptoms, disability, and financial impacts, measured repeatedly over 36 months.

ELIGIBILITY:
Inclusion Criteria:

* All VA enrollees since February 2020, which includes all patients who were tested for SARS-CoV-2 and are included in the VA COVID-19 Shared Data Resource in CDW.

Exclusion Criteria:

* VA employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All VA enrollees since February 2020, which includes all patients who were tested for SARS-CoV-2 and are included in the VA COVID-19 Shared Data Resource in CDW.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise M. Hynes, PhD MPH RN, Principal Investigator — VA Portland Health Care System, Portland, OR; Matthew L Maciejewski, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Amy S Bohnert, PhD MHS BA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Elizabeth M Viglianti, MD MPH MSc, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Ann M. O'Hare, MD MA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; George N. Ioannou, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (6):
- United States (6):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Beginning six months after the first survey is collected, updated releases of all structured survey items and basic summary scores will be released via VINCI for all VA investigators with appropriate permissions-but specific HIPAA-protected identifiers will not be included. The research information sheet and recruitment letter include the VA's recommended explicit language about this and the option to opt out.
Supporting Information: Study Protocol
Time Frame: Releases of survey items and scores will occur every six months and will be available indefinitely
Access Criteria: Researchers that access this data for future research use may be national or international and affiliated or unaffiliated with the VA, and may only use the data for research purposes. Future studies will have appropriate data use agreements in place as well as receive approval by an IRB and other oversight committees prior to starting any research.

REFERENCES:
- [Background] Ioannou GN, Ferguson JM, O'Hare AM, Bohnert ASB, Backus LI, Boyko EJ, Osborne TF, Maciejewski ML, Bowling CB, Hynes DM, Iwashyna TJ, Saysana M, Green P, Berry K. Changes in the associations of race and rurality with SARS-CoV-2 infection, mortality, and case fatality in the United States from February 2020 to March 2021: A population-based cohort study. PLoS Med. 2021 Oct 21;18(10):e1003807. doi: 10.1371/journal.pmed.1003807. eCollection 2021 Oct. PMID 34673772
- [Result] Ioannou GN, Bohnert ASB, O'Hare AM, Boyko EJ, Maciejewski ML, Smith VA, Bowling CB, Viglianti E, Iwashyna TJ, Hynes DM, Berry K; COVID-19 Observational Research Collaboratory (CORC). Effectiveness of mRNA COVID-19 Vaccine Boosters Against Infection, Hospitalization, and Death: A Target Trial Emulation in the Omicron (B.1.1.529) Variant Era. Ann Intern Med. 2022 Dec;175(12):1693-1706. doi: 10.7326/M22-1856. Epub 2022 Oct 11. PMID 36215715
- [Result] O'Hare AM, Vig EK, Iwashyna TJ, Fox A, Taylor JS, Viglianti EM, Butler CR, Vranas KC, Helfand M, Tuepker A, Nugent SM, Winchell KA, Laundry RJ, Bowling CB, Hynes DM, Maciejewski ML, Bohnert ASB, Locke ER, Boyko EJ, Ioannou GN; VA COVID Observational Research Collaboratory (CORC). Complexity and Challenges of the Clinical Diagnosis and Management of Long COVID. JAMA Netw Open. 2022 Nov 1;5(11):e2240332. doi: 10.1001/jamanetworkopen.2022.40332. PMID 36326761
- [Result] Bajema KL, Wang XQ, Hynes DM, Rowneki M, Hickok A, Cunningham F, Bohnert A, Boyko EJ, Iwashyna TJ, Maciejewski ML, Viglianti EM, Streja E, Yan L, Aslan M, Huang GD, Ioannou GN. Early Adoption of Anti-SARS-CoV-2 Pharmacotherapies Among US Veterans With Mild to Moderate COVID-19, January and February 2022. JAMA Netw Open. 2022 Nov 1;5(11):e2241434. doi: 10.1001/jamanetworkopen.2022.41434. PMID 36367727
- [Result] Admon AJ, Wander PL, Iwashyna TJ, Ioannou GN, Boyko EJ, Hynes DM, Bowling CB, Bohnert ASB, O'Hare AM, Smith VA, Pura J, Hebert PL, Wong ES, Niederhausen M, Maciejewski ML. Consensus elements for observational research on COVID-19-related long-term outcomes. Medicine (Baltimore). 2022 Nov 18;101(46):e31248. doi: 10.1097/MD.0000000000031248. PMID 36401423
- [Result] Bajema KL, Rowneki M, Berry K, Bohnert A, Bowling CB, Boyko EJ, Iwashyna TJ, Maciejewski ML, O'Hare AM, Osborne TF, Viglianti EM, Hynes DM, Ioannou GN. Rates of and Factors Associated With Primary and Booster COVID-19 Vaccine Receipt by US Veterans, December 2020 to June 2022. JAMA Netw Open. 2023 Feb 1;6(2):e2254387. doi: 10.1001/jamanetworkopen.2022.54387. PMID 36729454
- [Result] Bohnert AS, Kumbier K, Rowneki M, Gupta A, Bajema K, Hynes DM, Viglianti E, O'Hare AM, Osborne T, Boyko EJ, Young-Xu Y, Iwashyna TJ, Maciejewski M, Schildhouse R, Dimcheff D, Ioannou GN. Adverse outcomes of SARS-CoV-2 infection with delta and omicron variants in vaccinated versus unvaccinated US veterans: retrospective cohort study. BMJ. 2023 May 23;381:e074521. doi: 10.1136/bmj-2022-074521. PMID 37220941
- [Result] Smith VA, Berkowitz TSZ, Hebert P, Wong ES, Niederhausen M, Pura JA, Berry K, Green P, Korpak A, Fox A, Baraff A, Hickok A, Shahoumian TA, Bohnert ASB, Hynes DM, Boyko EJ, Ioannou GN, Iwashyna TJ, Bowling CB, O'Hare AM, Maciejewski ML. Correction: Design and analysis of outcomes following SARS-CoV-2 infection in veterans. BMC Med Res Methodol. 2023 Aug 25;23(1):194. doi: 10.1186/s12874-023-02021-4. No abstract available. PMID 37620765
- [Result] Hynes DM, Niederhausen M, Chen JI, Shahoumian TA, Rowneki M, Hickok A, Shepherd-Banigan M, Hawkins EJ, Naylor J, Teo A, Govier DJ, Berry K, McCready H, Osborne TF, Wong E, Hebert PL, Smith VA, Bowling CB, Boyko EJ, Ioannou GN, Iwashyna TJ, Maciejewski ML, O'Hare AM, Viglianti EM, Bohnert AS. Risk of Suicide-Related Outcomes After SARS-COV-2 Infection: Results from a Nationwide Observational Matched Cohort of US Veterans. J Gen Intern Med. 2024 Mar;39(4):626-635. doi: 10.1007/s11606-023-08440-9. Epub 2023 Oct 26. PMID 37884839
- [Result] Ioannou GN, Berry K, Rajeevan N, Li Y, Mutalik P, Yan L, Bui D, Cunningham F, Hynes DM, Rowneki M, Bohnert A, Boyko EJ, Iwashyna TJ, Maciejewski ML, Osborne TF, Viglianti EM, Aslan M, Huang GD, Bajema KL. Effectiveness of Nirmatrelvir-Ritonavir Against the Development of Post-COVID-19 Conditions Among U.S. Veterans : A Target Trial Emulation. Ann Intern Med. 2023 Nov;176(11):1486-1497. doi: 10.7326/M23-1394. Epub 2023 Oct 31. PMID 37903369
- [Result] Wander PL, Baraff A, Fox A, Cho K, Maripuri M, Honerlaw JP, Ho YL, Dey AT, O'Hare AM, Bohnert ASB, Boyko EJ, Maciejewski ML, Viglianti E, Iwashyna TJ, Hynes DM, Osborne TF, Ioannou GN. Rates of ICD-10 Code U09.9 Documentation and Clinical Characteristics of VA Patients With Post-COVID-19 Condition. JAMA Netw Open. 2023 Dec 1;6(12):e2346783. doi: 10.1001/jamanetworkopen.2023.46783. PMID 38064215
- [Result] Hebert PL, Kumbier KE, Smith VA, Hynes DM, Govier DJ, Wong E, Kaufman BG, Shepherd-Banigan M, Rowneki M, Bohnert ASB, Ioannou GN, Boyko EJ, Iwashyna TJ, O'Hare AM, Bowling CB, Viglianti EM, Maciejewski ML; VA COVID-19 Observational Research Collaboratory (CORC). Changes in Outpatient Health Care Use After COVID-19 Infection Among Veterans. JAMA Netw Open. 2024 Feb 5;7(2):e2355387. doi: 10.1001/jamanetworkopen.2023.55387. PMID 38334995
- [Result] Iwashyna TJ, Seelye S, Berkowitz TS, Pura J, Bohnert ASB, Bowling CB, Boyko EJ, Hynes DM, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Womer J, Prescott HC, Smith VA; VA HSR&D COVID-19 Observational Research Collaboratory. Late Mortality After COVID-19 Infection Among US Veterans vs Risk-Matched Comparators: A 2-Year Cohort Analysis. JAMA Intern Med. 2023 Oct 1;183(10):1111-1119. doi: 10.1001/jamainternmed.2023.3587. PMID 37603339
- [Result] Iwashyna TJ, Smith VA, Seelye S, Bohnert ASB, Boyko EJ, Hynes DM, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Berkowitz TS, Pura J, Womer J, Kamphuis LA, Monahan ML, Bowling CB; VA HSR&D COVID-19 Observational Research Collaboratory (CORC). Self-Reported Everyday Functioning After COVID-19 Infection. JAMA Netw Open. 2024 Mar 4;7(3):e240869. doi: 10.1001/jamanetworkopen.2024.0869. PMID 38427352
- [Result] Ioannou GN, Baraff A, Fox A, Shahoumian T, Hickok A, O'Hare AM, Bohnert ASB, Boyko EJ, Maciejewski ML, Bowling CB, Viglianti E, Iwashyna TJ, Hynes DM. Rates and Factors Associated With Documentation of Diagnostic Codes for Long COVID in the National Veterans Affairs Health Care System. JAMA Netw Open. 2022 Jul 1;5(7):e2224359. doi: 10.1001/jamanetworkopen.2022.24359. PMID 35904783
- [Result] Chen JI, Bui D, Iwashyna TJ, Shahoumian TA, Hickok A, Shepherd-Banigan M, Hawkins EJ, Naylor J, Govier DJ, Osborne TF, Smith VA, Bowling CB, Boyko EJ, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Bohnert AS, Hynes DM; V. A. HSRDSARS-C.O.V.-2 Observational Research Collaboratory (CORC). Impact of SARS-CoV-2 Infection on Long-Term Depression Symptoms among Veterans. J Gen Intern Med. 2024 Jun;39(8):1310-1316. doi: 10.1007/s11606-024-08630-z. Epub 2024 Apr 16. PMID 38625482
- [Result] Chen JI, Bui D, Iwashyna TJ, Shahoumian TA, Hickok A, Shepherd-Banigan M, Hawkins EJ, Naylor J, Govier DJ, Osborne TF, Smith VA, Bowling CB, Boyko EJ, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Bohnert AS, Hynes DM; V. A. HSRDSARS-C.O.V.-2 Observational Research Collaboratory (CORC). Correction to: Impact of SARS-CoV-2 Infection on Long-Term Depression Symptoms among Veterans. J Gen Intern Med. 2024 May 14. doi: 10.1007/s11606-024-08800-z. Online ahead of print. No abstract available. PMID 38743168
- [Result] Hauschildt KE, Bui DP, Govier DJ, Eaton TL, Viglianti EM, Ettman CK, McCready H, Smith VA, O'Hare AM, Osborne TF, Boyko EJ, Ioannou GN, Maciejewski ML, Bohnert ASB, Hynes DM, Iwashyna TJ; VA COVID-19 Observational Research Collaboratory (CORC). Regional variation in financial hardship among US veterans during the COVID-19 pandemic. Health Aff Sch. 2024 Jun 5;2(6):qxae075. doi: 10.1093/haschl/qxae075. eCollection 2024 Jun. PMID 38938272
- [Result] Govier DJ, Bui DP, Hauschildt KE, Eaton TL, McCready H, Smith VA, Osborne TF, Bowling CB, Boyko EJ, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Bohnert ASB, Hynes DM, Iwashyna TJ. Financial hardship after COVID-19 infection among US Veterans: a national prospective cohort study. BMC Health Serv Res. 2024 Aug 19;24(1):943. doi: 10.1186/s12913-024-11421-1. PMID 39160528
- [Result] Ioannou GN, Berry K, Rajeevan N, Li Y, Yan L, Huang Y, Lin HM, Bui D, Hynes DM, Rowneki M, Bohnert A, Boyko EJ, Iwashyna TJ, Maciejewski ML, Smith VA, Berkowitz TSZ, O'Hare AM, Viglianti EM, Aslan M, Bajema KL. Effectiveness of the 2023-to-2024 XBB.1.5 COVID-19 Vaccines Over Long-Term Follow-up : A Target Trial Emulation. Ann Intern Med. 2025 Mar;178(3):348-359. doi: 10.7326/ANNALS-24-01015. Epub 2025 Feb 4. PMID 39903865
- [Result] Chen JI, Niederhausen M, Bui DP, Govier DJ, Rowneki M, Hickok A, Shahoumian TA, Shepherd-Banigan M, Korpak A, Hawkins E, Teo AR, Naylor J, Osborne TF, Smith VA, Bowling CB, Boyko EJ, Ioannou GN, Maciejewski ML, O'Hare AM, Viglianti EM, Iwashyna TJ, Bohnert ASB, Hynes DM; VA HSR&D COVID-19 Observational Research Collaboratory (CORC). Veteran Mental Health Emergency Care Utilization Following SARS-CoV-2 Infection. Health Serv Res. 2025 Oct;60(5):e14622. doi: 10.1111/1475-6773.14622. Epub 2025 Jun 5. PMID 40474431
- See also: VA COVID-19 Observational Research Collaboratory Website — https://www.research.va.gov/corc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We retrospectively assembled 14 monthly cohorts of Veterans with a first positive test for COVID-19 and up to 20 matched uninfected comparators between March 2020 and April 2021. Survey participants were sampled from this parent cohort. First, we randomly sampled 100 Veterans with COVID-19 from each month between Oct 2020 and April 2021. Sampled Veterans were invited to participate in surveys. If a sampled Veteran consented, we reached out to five of their matched comparators to participate.
Groups:
- Veterans Who Tested Positive for COVID-19 (Case): A random sample of Veterans who tested positive for COVID-19 between October 2020 and April 2021. The sampled Veterans who survived their initial SARS-CoV-2 infection were invited to participate in a series of four longitudinal surveys beginning approximately 18 months after their infection (or "index date"). After the first survey 18-month survey was completed, Veterans were contacted every 6-months to complete a follow-up survey up until 36-months after their initial infection or index date. In this arm, 235 consented and completed the initial survey and 220 completed all four surveys.
- Veterans Who Did Not Test Positive for COVID-19 (Comparator): To support causal inference, the investigators will also sample up to five comparator Veterans without COVID who are matched to participants with COVID-19 (within the same month of their infection). In general, cases will be compared to comparators matched on risk of developing COVID infection during a given wave. The five uninfected comparators were contacted after the matched index Veteran (case) consented to participate in surveys. The uninfected comparators were given the same series of surveys (four total beginning 18-months after their matched index date). In this arm, 244 consented and completed the initial survey and 220 completed all four.
Period: Overall Study
Arm/Group | Veterans Who Tested Positive for COVID-19 (Case) | Veterans Who Did Not Test Positive for COVID-19 (Comparator)
Started | 235 | 244
Completed | 220 | 220
Not Completed | 15 | 24

BASELINE CHARACTERISTICS:
Population: Baseline analysis included all Veterans who tested positive for COVID-19 and their matched comparators who consented to and responded to the first longitudinal survey cycle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Veterans Who Tested Positive for COVID-19 (Case) | Veterans Who Did Not Test Positive for COVID-19 (Comparator) | Total
Number analyzed (Participants) | 235 | 244 | 479
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [50 to 72] | 62 [48 to 72] | 61 [49 to 72]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 23 | 20 | 43
  Sex: Male | 183 | 124 | 307
  Sex: Unknown | 29 | 100 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 187 | 127 | 314
  Unknown or Not Reported | 34 | 101 | 135
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 48 | 36 | 84
  Race: White | 145 | 98 | 243
  Race: Other | 4 | 4 | 8
  Race: Unknown | 38 | 106 | 144
Region of Enrollment [Number; unit: participants]
  United States | 235 | 244 | 479
Baseline Instrumental Activities of Daily Living and Activities of Daily Living (I/ADL) [Count of Participants; unit: Participants] — Baseline Instrumental Activities and Activities of Daily Living (I/ADL) (18 months)
  Participants
    Difficulty dressing, including putting on shoes and socks: No | 161 | 178 | 339
    Difficulty dressing, including putting on shoes and socks: Yes | 63 | 57 | 120
    Difficulty dressing, including putting on shoes and socks: Don't do | 10 | 5 | 15
    Difficulty dressing, including putting on shoes and socks: Can't do | 0 | 0 | 0
    Difficulty dressing, including putting on shoes and socks: Unknown | 1 | 4 | 5
    Difficulty walking across room?: No | 171 | 177 | 348
    Difficulty walking across room?: Yes | 62 | 63 | 125
    Difficulty walking across room?: Don't do | 1 | 0 | 1
    Difficulty walking across room?: Can't do | 0 | 0 | 0
    Difficulty walking across room?: Unknown | 1 | 4 | 5
    Difficulty bathing or showering?: No | 185 | 191 | 376
    Difficulty bathing or showering?: Yes | 49 | 48 | 97
    Difficulty bathing or showering?: Don't do | 0 | 0 | 0
    Difficulty bathing or showering?: Can't do | 0 | 0 | 0
    Difficulty bathing or showering?: Unknown | 1 | 5 | 6
    Difficulty eating?: No | 219 | 224 | 443
    Difficulty eating?: Yes | 14 | 16 | 30
    Difficulty eating?: Don't do | 0 | 0 | 0
    Difficulty eating?: Can't do | 0 | 0 | 0
    Difficulty eating?: Unknown | 2 | 4 | 6
    Difficulty getting in or out of bed?: No | 168 | 172 | 340
    Difficulty getting in or out of bed?: Yes | 65 | 68 | 133
    Difficulty getting in or out of bed?: Don't do | 0 | 0 | 0
    Difficulty getting in or out of bed?: Can't do | 1 | 0 | 1
    Difficulty getting in or out of bed?: Unknown | 1 | 4 | 5
    Difficulty using toilet?: No | 184 | 196 | 380
    Difficulty using toilet?: Yes | 50 | 42 | 92
    Difficulty using toilet?: Don't do | 0 | 1 | 1
    Difficulty using toilet?: Can't do | 0 | 0 | 0
    Difficulty using toilet?: Unknown | 1 | 5 | 6
    Difficulty using map?: No | 199 | 217 | 416
    Difficulty using map?: Yes | 30 | 21 | 51
    Difficulty using map?: Don't do | 4 | 2 | 6
    Difficulty using map?: Can't do | 0 | 0 | 0
    Difficulty using map?: Unknown | 2 | 4 | 6
    Difficulty shopping for groceries?: No | 161 | 178 | 339
    Difficulty shopping for groceries?: Yes | 63 | 57 | 120
    Difficulty shopping for groceries?: Don't do | 10 | 5 | 15
    Difficulty shopping for groceries?: Can't do | 0 | 0 | 0
    Difficulty shopping for groceries?: Unknown | 1 | 4 | 5
    Difficulty preparing a hot meal?: No | 201 | 203 | 404
    Difficulty preparing a hot meal?: Yes | 24 | 32 | 56
    Difficulty preparing a hot meal?: Don't do | 9 | 5 | 14
    Difficulty preparing a hot meal?: Can't do | 0 | 0 | 0
    Difficulty preparing a hot meal?: Unknown | 1 | 4 | 5
    Difficulty making phone calls?: No | 209 | 226 | 435
    Difficulty making phone calls?: Yes | 25 | 14 | 39
    Difficulty making phone calls?: Don't do | 0 | 0 | 0
    Difficulty making phone calls?: Can't do | 0 | 0 | 0
    Difficulty making phone calls?: Unknown | 1 | 4 | 5
    Difficulty making medications?: No | 188 | 208 | 396
    Difficulty making medications?: Yes | 42 | 30 | 72
    Difficulty making medications?: Don't do | 4 | 1 | 5
    Difficulty making medications?: Can't do | 0 | 0 | 0
    Difficulty making medications?: Unknown | 1 | 5 | 6
    Difficulty managing money?: No | 180 | 200 | 380
    Difficulty managing money?: Yes | 48 | 35 | 83
    Difficulty managing money?: Don't do | 6 | 5 | 11
    Difficulty managing money?: Can't do | 0 | 0 | 0
    Difficulty managing money?: Unknown | 1 | 4 | 5
    Difficulty stooping or kneeling?: No | 63 | 81 | 144
    Difficulty stooping or kneeling?: Yes | 166 | 155 | 321
    Difficulty stooping or kneeling?: Don't do | 2 | 0 | 2
    Difficulty stooping or kneeling?: Can't do | 3 | 3 | 6
    Difficulty stooping or kneeling?: Unknown | 1 | 5 | 6
    Difficulty lifting over 10 pounds?: No | 135 | 138 | 273
    Difficulty lifting over 10 pounds?: Yes | 93 | 100 | 193
    Difficulty lifting over 10 pounds?: Don't do | 1 | 2 | 3
    Difficulty lifting over 10 pounds?: Can't do | 5 | 0 | 5
    Difficulty lifting over 10 pounds?: Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Instrumental Activities of Daily Living and Activities of Daily Living (I/ADL) Score
Description: Measures level of disability on a scale from 0 - 14, where higher values are considered a worse outcome. Multiple survey timepoints will allow us to assess change in disability over time. The score consists of 14 questions about activities of daily living. The I/ADL score is a sum total of reported limitations ranging from 0 (no limitations reported) to 14 (limitations in all activities asked reported).
Time Frame: Survey months 18, 24, 30, 36
Measure: Mean (Standard Deviation); unit: I/ADL Score
Arm/Group | Veterans Who Tested Positive for COVID-19 (Case) | Veterans Who Did Not Test Positive for COVID-19 (Comparator)
Number analyzed (Participants) | 235 | 244
I/ADL Score
  18-month I/ADL Score | 3.40 (3.18) | 3.05 (3.09)
  24-month I/ADL Score | 3.50 (3.40) | 3.40 (3.30)
  30-month I/ADL Score | 3.31 (3.39) | 2.98 (2.88)
  36-month I/ADL Score | 3.60 (3.50) | 3.30 (3.20)
Statistical Analysis 1: Comparison: Veterans Who Tested Positive for COVID-19 (Case) vs Veterans Who Did Not Test Positive for COVID-19 (Comparator); Null hypothesis no difference in trends of I/ADL scores between Veterans with COVID-19 and comparators. We used adjusted linear mixed model (LMM) to model ADL scores over time (i.e., survey cycles) and by COVID-19 status. The LMM included an interaction term for time and COVID-19 status. LMM models were fitted with random intercepts (i.e., patient ID) and slopes (i.e., survey cycle). LMMs included fixed effects for patient baseline age, sex, and care assessment needs score; Test type: Superiority; p = 0.77, likelihood ratio test; Interaction = 0.02, 95% CI 2-sided [-0.13 to 0.18] — Beta for time by COVID-19 status
Statistical Analysis 2: Comparison: Veterans Who Tested Positive for COVID-19 (Case); Null hypothesis no difference in trends of I/ADL scores between Veterans with COVID-19 and comparators. We used adjusted linear mixed model (LMM) to model I/ADL scores over time (i.e., survey cycles) and by COVID-19 status. The LMM included an interaction term for time and COVID-19 status. LMM models were fitted with random intercepts (i.e., patient ID) and slopes (i.e., survey cycle). LMMs included fixed effects for patient baseline age, sex, and care assessment needs score; Test type: Superiority; p = 0.60, likelihood ratio test; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.44 to 0.67] — Beta coefficient for mean difference in mean longitudinal I/ADL score

ADVERSE EVENTS:
Time Frame: 36 months
Description: No adverse events because this was a non interventional study
Arm/Group | Veterans Who Tested Positive for COVID-19 (Case) | Veterans Who Did Not Test Positive for COVID-19 (Comparator)
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/244
Serious Adverse Events (participants affected / at risk) | 0/235 | 0/244
Other Adverse Events (participants affected / at risk) | 0/235 | 0/244

LIMITATIONS AND CAVEATS:
While COVID-19 status was ascertained early in the pandemic through evidence of PCR test, we were unable to ascertain if uninfected comparators became infected over time due to uptake in home testing. This would have resulted in misclassification of the uninfected and biased our results towards the null.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT05394025/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT05394025/SAP_002.pdf
  • Informed Consent Form (2022-07-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT05394025/ICF_000.pdf